CLINICAL TRIAL: NCT01957267
Title: Longitudinal Observational Study Using Functional and Structural Optical Coherence Tomography to Diagnose and Guide Treatment of Glaucoma
Brief Title: Functional and Structural Imaging for Glaucoma
Acronym: FSOCT
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Aiyin Chen, MD, Professor of Ophthalmology, Oregon Health & Science University, Oregon Health and Science University
Other Study IDs: OHSU IRB #00009729; 1R01EY023285 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-10-08 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
Keywords: Glaucoma; Optical Coherence Tomography; Intraocular pressure; Optic nervehead; Nerve fiber layer
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Glaucoma Group: Patients with clinically confirmed glaucomatous ONH or NFL defects, with or without VF abnormalities
- Normal Group: Volunteers with healthy eyes

SUMMARY:
The specific aims of the clinical studies are to:

* Develop a directional high-resolution OCT and OCT angiography prototype to improve imaging of structure and perfusion.
* Validate wide-field OCT and OCT angiography parameters to improve early glaucoma detection.
* Simulate visual field results by combining structural and angiography OCT data.
* Assess abilities of above technologies and OCT-derived parameters on predicting glaucoma detection, conversion, and progression.

DETAILED DESCRIPTION:
Glaucoma is the second leading cause of blindness in the US. The diagnosis and monitoring of glaucoma are important problems, not only because of its prevalence, but also because of its silent and irreversible nature. However all of the current diagnostic tests have serious limitations. Although elevated intraocular pressure (IOP) is a risk factor, most glaucoma patients actually have IOP within normal range. Visual field (VF) tests are poorly reproducible, and a series of 3 tests are needed to establish diagnosis or confirm progression. Although ophthalmoscopic examination can detect optic nerve head (ONH) and nerve fiber layer (NFL) defects, reliability in diagnosis and tracking is hampered by its subjective and semi-quantitative nature. Although quantitative imaging with optical coherence tomography (OCT), scanning laser polarimetry (SLP), and confocal scanning laser ophthalmoscopy (cSLO) can more objectively detect ONH and NFL defects, their diagnostic accuracies are still not sufficient to be relied on alone for diagnostic screening. It has been estimated that about half of glaucoma patients in the US do not know that they have the disease. Thus, there is a need for improvements in glaucoma diagnostic technologies. One approach that deserves further exploration is blood flow imaging.

There is much circumstantial evidence that vascular factors play important roles in the pathophysiology of glaucoma:

1. Systemic vasculopathy increases the risk of developing glaucoma. Hypertension, diabetes, and vasospastic conditions are all known risk factors. Normal tension glaucoma has also been linked to peripheral endothelial dysfunction and erectile dysfunction. This suggests that poor circulation may be a causative factor or a facilitative factor that predisposes the ONH to damage by elevated IOP.
2. Decrease or fluctuation in ocular perfusion pressure was identified as an independent risk factor for progression in the Collaborative Normal-Tension Glaucoma Study and other studies. Nocturnal hypotension is also a risk factor for glaucoma progression.
3. Medications that improve ocular perfusion appear to have protective effects that are not explained by the lowering of IOP.
4. Optic disc hemorrhage and peripapillary atrophy are both associated with accelerated glaucoma progression. These finding may support a role for focal ischemia.
5. Animal experiments show that increased IOP causes decreased ONH blood flow in the presence of low systemic blood pressure.

Despite the evidence, the management of glaucoma remains focused on the lowering of IOP, the one causative factor that responds to treatment and can be easily measured. Blood flow measurement is a research topic, but currently has no clinical role in the diagnosis, prognostic evaluation, or treatment of glaucoma. Therapies aimed at improving ocular circulation cannot be effectively developed without a practical method for quantitative and reproducible evaluation of ONH and retinal perfusion. Thus there is a great need to develop better technology for the evaluation of ocular circulation.

Using high-speed OCT systems, we have developed new methods to image and measure optic nerve head (ONH) and retinal blood flow. Preliminary results showed that VF loss was more highly correlated with retinal blood flow as measured by OCT than any neural structure measured by OCT or other imaging modality. Accordingly, the goal of the proposed project is to improve the diagnostic and prognostic evaluation of glaucoma by further developing novel functional OCT measurements using ultrahigh-speed (70-100 kHz) OCT technology.

Retinal blood flow, ONH circulation, optic disc rim volume, peripapillary nerve fiber layer volume, and macular ganglion cell complex volume are all pieces of the same glaucoma puzzle. This project will develop novel imaging methods that allow us to look at the whole picture using one tool - ultrahigh-speed OCT.

ELIGIBILITY:
Inclusion Criteria: Normal Subjects (both eyes must meet all criteria)

1. No history or evidence of retinal pathology or glaucoma
2. Normal Humphrey 24-2 VF: A mean defect (MD), corrected pattern standard deviation (CPSD) within 95% limits of normal reference, and glaucoma hemifield test (GHT) within normal limits (97%).
3. Intraocular pressure < 21 mm Hg
4. Central corneal pachymetry > 500 microns
5. No chronic ocular or systemic corticosteroid use
6. Open angle (gonioscopy must show 75% or more of the angle to be Grade 2 or more by Shaffer's grading system)
7. Normal appearing ONH and NFL: vertical and horizontal cup/disc ratio (CDR) ≤ 0.5 and intact neuroretinal rim without peripapillary hemorrhages, notches, localized pallor, or NFL defect
8. Symmetric ONH between left and right eyes: CDR difference < 0.2 in both vertical and horizontal dimensions

Inclusion criteria: Glaucoma Group

1. ONH or NFL defect visible on slit-lamp biomicroscopy defined as one of following:

   1. diffuse or localized thinning of the rim
   2. disc (splinter) hemorrhage
   3. notch in the rim
   4. vertical cup/disc ratio greater than the fellow eye by > 0.2
2. Presence or absence of VF defects as measured by Humphrey SITA 24-2 VF.

Exclusion Criteria: All Groups

1. Best-corrected visual acuity less than 20/40
2. Age < 40 or >85 years
3. Refractive error of > +3.00 D or < -7.00 D
4. Previous intraocular surgery except for uncomplicated keratorefractive surgery and cataract extraction with posterior chamber intraocular lens implantation
5. Diabetic retinopathy
6. Other diseases that may cause VF loss or optic disc abnormalities
7. Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil
8. Inability to perform reliably on automated VF testing
9. Life-threatening or debilitating illness making it unlikely patient could successfully complete the study.
10. Refusal of informed consent or of commitment to the full length of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll both males and females and include all ethnic and racial groups through clinical practices in the centers. The study will enroll subjects in the older adult age range commonly affected by glaucoma - 40 years or older. The study will exclude people with life-threatening or debilitating illness that would make 5-year participation unlikely or cooperation with tests difficult. For similar reasons those older than 85 years are excluded. The study also excludes those with any disease that might confound the diagnosis of glaucoma. Otherwise people with any health status are eligible for enrollment. Two groups of participants are recruited in the study: healthy controls or participants with confirmed glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-09-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Measure of retinal non-perfusion areas in mm2 | 5 years
Measure vessel density in percentage (%) | 5 years
Determine accuracy of sector visual field progression in OCT-based sector visual field simulation compared to actual visual field results. Measured in dB change over time. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aiyin Chen, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Casey Eye Institute, Portland, Oregon, United States